CLINICAL TRIAL: NCT02265679
Title: A Randomized, Double-blind Within Dose, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of Increasing Single Oral Doses of BIIL 284 BS in Adult and Pediatric Cystic Fibrosis Patients
Brief Title: Safety, Tolerability and Pharmacokinetics of Increasing Doses of BIIL 284 BS in Adult and Pediatric Cystic Fibrosis (CF) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 543.36
Record Dates: First submitted 2014-10-15; First posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — amelubant

ARMS (7):
- BIIL 284 BS, low dose in pediatric patients (Experimental)
  Interventions: Drug: BIIL 284 BS, low dose, pediatric patients
- BIIL 284 BS, medium dose in pediatric patients (Experimental)
  Interventions: Drug: BIIL 284 BS, medium dose, pediatric patients
- BIIL 284 BS, high dose in pediatric patients (Experimental)
  Interventions: Drug: BIIL 284 BS, high dose, pediatric patients
- BIIL 284 BS, low dose in adult patients (Experimental)
  Interventions: Drug: BIIL 284 BS, low dose, adult patients
- BIIL 284 BS, medium dose in adult patients (Experimental)
  Interventions: Drug: BIIL 284 BS, medium dose, adult patients
- BIIL 284 BS, high dose in adult patients (Experimental)
  Interventions: Drug: BIIL 284 BS, high dose, adult patients
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIL 284 BS, low dose, pediatric patients
  Arms: BIIL 284 BS, low dose in pediatric patients
Drug: BIIL 284 BS, medium dose, pediatric patients
  Arms: BIIL 284 BS, medium dose in pediatric patients
Drug: BIIL 284 BS, high dose, pediatric patients
  Arms: BIIL 284 BS, high dose in pediatric patients
Drug: BIIL 284 BS, low dose, adult patients
  Arms: BIIL 284 BS, low dose in adult patients
Drug: BIIL 284 BS, medium dose, adult patients
  Arms: BIIL 284 BS, medium dose in adult patients
Drug: BIIL 284 BS, high dose, adult patients
  Arms: BIIL 284 BS, high dose in adult patients
Drug: Placebo
  Arms: Placebo

SUMMARY:
Safety, tolerability and pharmacokinetics following single doses

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study were cystic fibrosis patients:
* Male or female ≥6 years (pediatrics 6 - 17 years; adult ≥18 years); minimum weight requirement of 20 kg
* Confirmed diagnosis of CF (positive sweat chloride ≥60 milliequivalents (mEq)/liter (by pilocarpine iontophoresis) and/or a genotype with two identifiable mutations consistent with CF accompanied by one or more clinical features with the CF phenotype
* Forced expiratory volume in one second (FEV1) >25% predicted (using prediction equation's of Knudson)
* Clinically stable with no evidence of acute upper or lower respiratory tract infection or current pulmonary exacerbation within 2 weeks of screening
* Females of child bearing potential needed to have a negative pregnancy test at screening and, if sexually active, had to be willing to use a double-barrier form of contraception for the duration of the study
* The patient or the patient's legally acceptable representative had to be able to give informed consent in accordance with international conference of harmonization (ICH) good clinical practice (GCP) guidelines and local legislation
* The patient must be able to swallow the BIIL 284 BS tablet whole
* Patients taking a chronic medication must be willing to continue this therapy for the entire duration of the study

Exclusion Criteria:

* Patients with a history of allergy/hypersensitivity (including medication allergy) which is deemed relevant to the trial as judged by the Investigator
* Patients who had participated in another study with an investigational drug within one month or 6 half-lives (whichever is greater) preceding the screening visit
* Patients with known substance abuse, including alcohol or drug abuse, within 30 days prior to screening
* Patients who participated in excessive physical activities (e.g. strenuous sporting events) within 24 hours before the study
* Female patients who were pregnant or lactating
* Patients who were unable to comply with breakfast requirements prior to dosing
* Patients who had received IV, oral or inhaled antibiotics or corticosteroids for a pulmonary exacerbation within 2 weeks of screening
* Patients who had started a new chronic medication for CF within 2 weeks of screening
* Patients with documented persistent colonization with B. cepacia (defined as more than one positive culture within the past year)
* Patients with clinically significant findings on chest x-ray which in the opinion of the Investigator precludes the patient's participation in the trial
* Patients with oxyhemoglobin saturation in room air <90% by pulse oximetry
* Patients with hemoglobin <9.0 g/dL; platelets <100x109/L; serum glutamic-oxaloacetic transaminase (ALT) or serum glutamic-pyruvic transaminase (AST) >2 times the upper limit of normal; creatinine >1.8 mg/dL at screening
* Clinically significant disease or medical condition other than CF or CF-related conditions that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data. This includes significant hematological, hepatic, renal, cardiovascular, and neurologic disease. Patients with diabetes may participate if their disease is under good control prior to screening.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2001-10; Primary Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in physical examination | Pre-dose and up to 5 days after drug administration
Number of patients with clinically relevant changes in vital signs (blood pressure, pulse rate, respiratory rate, body temperature) | Pre-dose, up to 5 days after drug administration
Changes from baseline in spirometry | Pre-dose and up to 5 days after drug administration
Changes from baseline in oximetry | Pre-dose and up to 5 days after drug administration
Number of patients with clinically relevant changes in 12-lead ECG | Pre-dose, up to 5 days after drug administration
Number of patients with clinically relevant changes in laboratory evaluation | Pre-dose, up to 5 days after drug administration
Number of patients with adverse events | Up to 5 days after drug administration

SECONDARY OUTCOMES:
Plasma concentration-time profiles of BIIL 315 ZW in all dose groups | Up to 5 days after drug administration
Plasma concentration-time profiles of BIIL 284 BS, BIIL 260 BS and BIIL 304 ZW in medium dose adult and high dose pediatric group | Up to 5 days after drug administration
Area under the concentration-time curve of the analytes in plasma (AUC) | Up to 5 days after drug administration
Maximum measured concentration of the analytes in plasma (Cmax) | Up to 5 days after drug administration
Time from dosing to the maximum concentration of the analytes in plasma (tmax) | Up to 5 days after drug administration
Terminal half-life of the analytes in plasma (t1/2) | Up to 5 days after drug administration
Total mean residence time of the analytes in the body (MRTtot) | Up to 5 days after drug administration
Terminal rate constant of the analytes in plasma (λz) | Up to 5 days after drug administration
Apparent clearance of the analytes in plasma following extravascular administration (CL/F) | Up to 5 days after drug administration
Apparent volume of distribution during the terminal phase λz following extravascular administration (Vz/F) | Up to 5 days after drug administration